CLINICAL TRIAL: NCT00476437
Title: Safety and Effect of Biphasic Insulin Aspart 50 Compared to Biphasic Human Insulin 50 in Patients With Type 2 Diabetes Mellitus.
Brief Title: Safety and Effect of Biphasic Insulin Aspart 50 in Patients With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1864; JapicCTI-070408 (Registry Identifier: japic)
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: biphasic human insulin

SUMMARY:
This trial is conducted in Japan. The purpose of this trial is to investigate the safety and the effect of biphasic insulin aspart 50 compared to biphasic human insulin 50 in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Current treatment with pre-mixed human insulin preparation or biphasic/pre-mixed insulin analogue in twice daily treatment for at least 8 weeks.
* HbA1C: less than 11.0%
* BMI: less than 30.0 kg/m2

Exclusion Criteria:

* Total daily insulin dose: 100 IU/U and more
* Treatment with oral hypoglycaemic agents within the last 4 weeks.
* Treatment with insulin sensitizer within the last 12 weeks
* A lifestyle that is considered unsuitable for this trial (frequent or routine night shift workers etc.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoglycaemic episodes | During 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com